CLINICAL TRIAL: NCT00411606
Title: Normal Values of Facial Thermography
Status: Completed | Type: Observational
Sponsor: West Penn Allegheny Health System (Other)
Collaborators: Greer Laboratories (Industry)
Responsible Party: David Skoner/Principal Investigator, Allegheny General Hospital
Other Study IDs: RC - 4220
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Healthy; Allergy; Allergic Rhinoconjunctivitis
Keywords: Healthy; Allergy; Allergic Rhinoconjunctivitis
MeSH Terms: conditions — Hypersensitivity | interventions — Thermography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Subjects with no allergies
  Interventions: Procedure: Thermography

INTERVENTIONS:
Procedure: Thermography — Subjects will have a picture of their face taken with a thermal camera

SUMMARY:
An objective of this study is to standardize temperature values derived from thermograms of the facial region. It is anticipated that the mean temperature of a defined region of interest, such as the eyes, nose, or sinuses, might be useful for future applications.

The investigators will attempt to determine normal temperature ranges based on participants' age and gender.

DETAILED DESCRIPTION:
Medical thermography is a noninvasive technique that allows an examiner to visualize and estimate the temperature of the skin surface. An infrared scanning device is used to convert infrared radiation emitted from the skin surface into electrical impulses that can be captured as an image called a thermogram. During the past 20 years medical thermography has been used to study the pathology in the vascular, muscular, neural and skeletal systems.

An objective of this study is to standardize temperature values derived from thermograms of the facial region. It is anticipated that the mean temperature of a defined region of interest, such as the eyes, nose, or sinuses, might be useful for future applications. This protocol addresses the definition of overall health, symptomology, and anthropometrical features (age, weight, height, body mass index and gender), and what effect, if any, each has on mean temperature. Environmental conditions, mapping procedures, and image evaluations will also be standardized. We will attempt to determine normal temperature ranges based on participants' age and gender. Future use of standardized values will be to assess the severity of rhinoconjunctivitis symptoms being experienced by a subject.

Subjects will make one visit to our clinic. They will be asked to acclimate to room temperature for at least 30 minutes. Subjects are requested not to consume hot drinks or food for at least an hour before imaging and not to use any skin preparations such as creams or talcum powder. A picture of the participant's face will be taken using the thermal camera which will demonstrate the temperature of each facial area of interest.

Please note that participants in this study will take part on a completely voluntary basis. No payment will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 7 and 70
* No mobility problems
* No restrictions in performing normal activities
* No regular pain or discomfort
* No anxiety or depression

Exclusion Criteria:

* Restrictions in performing normal activities
* Regular pain
* Anxiety or Depression
* Mobility problems

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: outpatient subjects at Allegheny General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoner, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States